CLINICAL TRIAL: NCT01653613
Title: Genomic Analysis of Adolescent and Young Adult Acute Lymphoblastic Leukemia
Brief Title: Studying Genes in Samples From Younger Patients With Acute Lymphoblastic Leukemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Robert L. Comis, ECOG Group Chair's Office
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: ECOG-E2L10T1; CDR0000737435 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Leukemia
Keywords: B-cell adult acute lymphoblastic leukemia; B-cell childhood acute lymphoblastic leukemia; untreated adult acute lymphoblastic leukemia; untreated childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia | interventions — In Situ Hybridization, Fluorescence; Gene Expression Profiling; Microarray Analysis; Amplified Fragment Length Polymorphism Analysis; Reverse Transcriptase Polymerase Chain Reaction

INTERVENTIONS:
Genetic: DNA analysis
Genetic: fluorescence in situ hybridization
Genetic: gene expression analysis
Genetic: microarray analysis
Genetic: mutation analysis
Genetic: polymorphism analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and bone marrow from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors find better ways to treat cancer.

PURPOSE: This laboratory study is looking into genes in samples from younger patients with acute lymphoblastic leukemia (ALL).

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify somatically acquired genetic copy number and sequence alterations at the time of diagnosis in adolescent and young adults (AYA) acute lymphoblastic leukemia (ALL) samples and to correlate them with clinical and laboratory characteristics and outcome.
* To identify specific microarray multi-gene and multi-exon expression signatures at the time of diagnosis and to correlate them with clinical and laboratory characteristics and outcome.
* To gain insights into the genetic events that contribute to the formation, development and relapse of AYA ALL by integrating the copy number and sequence alterations with the multi-gene signatures and by comparing these with data already generated in pediatric ALL.

OUTLINE: Cryopreserved samples are analyzed for DNA copy number alterations and loss-of-heterozygosity, gene expression profiling, and mutation analysis by single nucleotide polymorphism (SNP) microarrays, Affymetrix Exon arrays, and whole genome amplification (WGA, Repli-G Qiagen). Confirmation studies are then done by fluorescence in situ hybridization (FISH), reverse transcriptase (RT)-polymerase chain reaction (PCR), and rapid amplification of cDNA ends (RACE).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Samples from patients diagnosed with B-progenitor AYA ALL from:

  * The Children's Oncology Group high risk ALL Study AALL0232 (age 16-21)
  * The St. Jude Children's Research Hospital (SJCRH) Total XV studies (age 16-21)
  * AYA ALL (from patients 22-30 years of age and from patients age 31-39 years) existing in the ALL Tissue Repositories of the adult National Cancer Institute (NCI) Cooperative Oncology Groups

    * The Cancer and Leukemia Group B (CALGB)
    * The Eastern Cooperative Oncology Group (ECOG)
    * The Southwest Oncology Group (SWOG)
* Cryopreserved viable leukemic cell suspensions, obtained from bone marrow or peripheral blood at pretreatment and initial diagnosis
* Matched normal (germline) samples from end induction-remission bone marrow or blood samples or from buccal swabs, if available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 16 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2010-08; Primary Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Identification of somatically acquired genetic copy number and sequence alterations
Associations between genetic lesions (including mutations and copy number alterations) and known prognostic factors such as age group and white blood count at the time of diagnosis group using a Fisher exact test or Chi squared
Association between genetic lesion and outcome using a Kaplan-Meier curve and perform logrank test for each lesion

CONTACTS AND LOCATIONS:
Overall Officials: Charles Mullighan, MD, Principal Investigator — St. Jude Children's Research Hospital